CLINICAL TRIAL: NCT06353334
Title: Butylphthalide's Safety and Efficacy for Improving Neurological Function Prognosis in Patients With Cardiac Arrest (BNCA Trial): A Single-Center, Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Butylphthalide's Safety and Efficacy for Improving Neurological Function Prognosis in Patients With Cardiac Arrest (BNCA Trial)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tang Ziren (Other)
Responsible Party: Sponsor-Investigator, Tang Ziren, Professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-3-22-8
Record Dates: First submitted 2024-04-02; First posted 2024-04-09 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Butylphthalide; Cardiac Arrest; Neuroprotective Drugs
MeSH Terms: conditions — Heart Arrest | interventions — 3-n-butylphthalide; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Butylphthalide (Experimental): Butylphthalide and Sodium Chloride Injection 100ml ivgtt bid 14days
  Interventions: Drug: Butylphthalide and Sodium Chloride Injection
- Saline Solution (Placebo Comparator): Saline Solution 100ml ivgtt bid 14days
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Butylphthalide and Sodium Chloride Injection — All enrolled patients will undergo standard treatment as per international guidelines, concurrently receiving either NBP or placebo therapy. Patients in the experimental group will receive intravenous infusion of 100ml NBP twice daily. Each patient will receive continuous medication for 14 days.
  Arms: Butylphthalide
Drug: Saline Solution — All enrolled patients will undergo standard treatment as per international guidelines, concurrently receiving either NBP or placebo therapy. Patients in the control group will receive intravenous infusion of 100ml saline solution twice daily. Each patient will receive continuous medication for 14 days.
  Arms: Saline Solution

SUMMARY:
Butylphthalide (NBP) is a neuroprotective medication capable of ameliorating neurological dysfunction induced by ischemia, hypoxia, and reperfusion injury in the brain. However, evidence regarding the improvement of neurological function prognosis in patients with return of spontaneous circulation (ROSC) after cardiac arrest (CA) by NBP is limited. This study aims to evaluate the safety and efficacy of NBP treatment in improving the neurological function prognosis of patients with ROSC after CA.The study will be a single-center, randomized, double-blind, placebo-controlled trial. The sample size is estimated to be 100 patients. Eligible patients will be randomly allocated in a 1:1 ratio to receive either NBP or placebo treatment daily for a duration of 14 days. The initial administration of NBP or placebo treatment will commence within 6 hours after ROSC following CA. The primary outcome is the proportion of patients with Cerebral Performance Category (CPC) scores of 1-2 at 90 days after randomization in each group. The primary safety outcome is the percentage of severe adverse events occurring during the 14-day treatment period. This trial will determine the efficacy of NBP in providing neuroprotective effects for patients with ROSC after CA.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old.
2. GCS scores ≤8 upon admission.
3. ROSC ≥30min.
4. Signed the informed consent form.

Exclusion Criteria:

1. Cardiac arrest due to irreversible causes such as trauma, poisoning, etc.
2. Cardiac arrest due to end-stage conditions such as advanced cancer.
3. Persistent cardiogenic shock that is unreversed (defined as a systolic blood pressure persistently <90mmHg despite treatment with fluid resuscitation, vasopressor agents, and inotropic medications).
4. Presence of pre-existing cerebrovascular disease prior to cardiac arrest or confirmed intracranial hemorrhage by CT scan following admission.
5. Pre-existing CPC scores of 3-5 prior to cardiac arrest.
6. Prior use of NBP or any medication containing NBP before cardiac arrest.
7. Presence of severe hepatic or renal dysfunction before cardiac arrest (defined as ≥3× upper limit of normal alanine transaminase or ≥2× upper limit of normal creatinine).
8. Bradycardia or sick sinus syndrome occurs after ROSC.
9. History of prior drug or food allergies, or known allergies to the medication components used in this study.
10. Existence of treatment limitations (patient or their legal representative refusing advanced life support treatment, including mechanical ventilation, chest compressions, targeted temperature management, etc.).
11. Presence of severe bleeding tendency upon admission.
12. Body temperature <30℃ upon admission.
13. Pregnant or lactating women, or reproductive-age females with elevated serum hCG levels.
14. Other conditions deemed unsuitable for this trial by the principal investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with a CPC score of 1-2 | 90 days
  The primary outcome is the proportion of patients with a CPC score of 1-2 at 90days after randomization in each group. Favourable: 1 means full recovery or mild disability, 2 means moderate disability but independent in activities of daily living (ADLs). Unfavourable: 3 means severe disability-Dependent in ADLs, 4 means persistent vegetive state, 5 means Death.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chao-Yang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 6 months after publication
Access Criteria: The de-identified survey data will be made available for research purposes by contacting the corresponding authors